CLINICAL TRIAL: NCT06225232
Title: An 8-week Phase 2 Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of Psilocybin-assisted-psychotherapy in Adults With Cannabis Use Disorder: A Proof-of-Concept Study
Brief Title: Psilocybin in the Treatment of Cannabis Use Disorder: A-Proof-of-Concept Study
Acronym: PSI_CUD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Center for Medicinal Cannabis Research (Other); Peter Boris Centre for Addictions Research (PBCAR) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSI_CUD
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-11

CONDITIONS: Cannabis Use Disorder, Moderate; Cannabis Use Disorder, Severe
Keywords: Cannabis Use Disorder; Psilocybin; Motivational Enhancement Therapy
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): This is an open-label single arm intervention trial. Participants in this arm will be offered both drug and psychotherapy as part of their 9-week intervention.
  Interventions: Drug: Psilocybin combined with Psychotherapy

INTERVENTIONS:
Drug: Psilocybin combined with Psychotherapy — The intervention consists of a 9-week treatment protocol that is based on supportive psychotherapy and Motivational Enhancement Therapy. Overall, the therapy course includes 8 motivational enhancement therapy sessions and two experimental drug sessions.

SUMMARY:
Cannabis is the most commonly used psychoactive substance in Canada (Lowry & Corsi, 2020). A sub-group of cannabis users develop a condition known as Cannabis Use Disorder (CUD), which is defined as a regular pattern of cannabis use that causes performance difficulty at work, school and relationships (Hasin et al., 2013). A review of current treatments available for CUD indicate the lack of a pharmacological and psychological treatment with high success rates, which highlights the importance of exploring potential psychosocial interventions for the treatment of CUD. Given the evidence of psilocybin's therapeutic potential in the treatment of substance use disorders (de Veen et al., 2017), we aim to conduct a study using psilocybin-assisted-psychotherapy in the treatment of CUD. The study aims to evaluate the feasibility, safety, tolerability and potential therapeutic effect of 2 doses [25 mg] of psilocybin administered as part of an 8-week Motivational Enhancement Therapy (MET) and supportive therapy. This trial will be the first to evaluate the potential treatment effects of psilocybin on symptoms of CUD.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form.
2. Able to show documentation of identity.
3. Fluent in speaking and reading English and able to complete rating scales and assessments.
4. Between the ages of 18 to 65.
5. At Screening, meet criteria for CUD diagnosis of at least moderate severity as per the MINI Plus
6. Expressed a wish to reduce or stop cannabis use.
7. Medically healthy based on physician review of CBC, electrolytes, liver function test, kidney function tests and ECG.
8. Has a stable residence for the duration of the study.
9. Agree to comply with the protocol requirements set out by the study.
10. Consent to providing regular check-ins and follow-up regarding any medical conditions, procedures and adverse events.
11. If of child-bearing potential, female participants must agree to use an adequate birth control method (IUD, injected or implanted hormonal methods, abstinence, vasectomy of the partner/partners, or double barrier contraception i.e. condoms plus diaphragm, or diaphragm plus spermicide) for the duration of the study. Male participants should agree to using condoms with spermicide throughout the trial in addition to the use of an adequate contraceptive by their partner of childbearing potential.
12. Following discharge from the dosing sessions, agree to have another individual accompany them home from the study site and stay with them overnight.

Exclusion Criteria:

1. Meet DSM-5 criteria for lifetime history of bipolar disorder, schizophrenia, or other psychotic disorders, personality disorders, delirium, dementia and amnesic and other cognitive disorders, or are in a current agitated state.
2. Have first-degree biological relatives (parents or full siblings) with past or present history of schizophrenia, bipolar disorder and any other psychosis.
3. Meet DSM-5 criteria for panic disorder or seizure disorders.
4. Meet DSM-5 criteria for dependence of any substance other than cannabis or tobacco in the past 6 months.
5. Positive urine drug screen for substances tested with the exception of cannabis
6. History of serotonergic psychedelic use in the past year and over 5 times of lifetime use (psilocybin, LSD, Ayahuasca, mescaline, DMT).
7. Current treatment with psychotropic agents including stimulants, anti-psychotic agents, benzodiazepines and tri-cyclic anti-depressants. Concurrent treatment with Selective Serotonin Reuptake Inhibitors and Serotonin Noradrenalin Reuptake Inhibitors will be allowed, provided the dose has been stable for 4 weeks and remains stable during the study.
8. History of cardiovascular diseases or uncontrolled hypertension that is not successfully treated or any other medical condition that might pose a risk to the participant in the opinion of the study physician.
9. Are receiving concurrent psychotherapy for CUD.
10. Are reasonably judged to present a serious suicide risk as determined by Columbia Suicide Severity Rating Scale or expressed homicide risk, who have enacted suicidal behaviors within 6 months prior to intake, or w ho are likely to require psychiatric hospitalization during the study.
11. Participants of childbearing potential with a positive pregnancy test at screening or prior to dosing sessions, or are pregnant, breast feeding, and who are not using an acceptable means of birth control for the duration of the study.
12. Are unable to fully understand the potential risks and benefits of the study and give informed consent.
13. Are currently or planning on participating in other interventional clinical trials during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of spontaneously reported adverse events and serious adverse events from baseline to the nine-week endpoint | 9 weeks
  frequency, type and severity of outcomes are recorded
Percent of recruited participants who discontinue or are lost to follow up before completing the 9-ween treatment protocol | 9 weeks
  frequency of cases of withdrawal and lost to follow up are documented and a percent is calculated based on the total number of participants recruited in this study.

SECONDARY OUTCOMES:
Feasibility measured by number of individuals who express interest by contacting the study team, percent of individuals who are screened as eligible to those who contact the study, percent of those who complete the trial to those who are enrolled | 9 weeks
  Reported in frequency and percentages
Efficacy a: frequency and amount of cannabis use, as measured by the Timeline Follow Back from baseline to the nine-week end point | 9 weeks
  This is measured using the Timeline Follow Back tool
Efficacy b: Severity of symptoms associated with Cannabis Use Disorder as measured by Self-Reported Symptoms of Cannabis Use Disorder from baseline to 9 week endpoint | 9 weeks
  Self-Reported Symptoms of Cannabis Use Disorder
Efficacy c: Changes in Urinary Cannabinoids from baseline to the nine-week endpoint | 9 weeks
  Urinary Cannabinoid Test

OTHER OUTCOMES:
severity of symptoms of craving, withdrawal, anxiety, depression and functional impairment | 9 weeks
  Measured using Marijuana Withdrawal Checklist, Marijuana Craving Questionnaire, Patient Health Questionnaire - 9, Generalized Anxiety Disorder, Sheehan Disability Scale

CONTACTS AND LOCATIONS:
Locations (1):
- MacAnxiety Research Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided